CLINICAL TRIAL: NCT05452889
Title: Utilizing 18F-fluoroglutamine PET Imaging in Patients With Pulmonary Arterial Hypertension
Brief Title: PET Image in PAH Patients
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Stephen Y. Chan (Other)
Collaborators: Bayer (Industry); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Stephen Y. Chan, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY21050035; PHAB Level 4 award 2021 (Other Grant/Funding Number: Bayer Healthcare Pharmaceuticals Inc.); R01HL124021 (NIH)
Record Dates: First submitted 2022-06-09; First posted 2022-07-11 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Pulmonary hypertension; Early diagnoses; Non invasive
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Hypertension, Pulmonary; Disease | interventions — N-(2-fluoropropionyl)glutamic acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 18F-FGLN PET Imaging (Experimental): 10.0 mCi of 18F-FGln will be injected intravenously as a slow bolus (20 sec)
  Interventions: Diagnostic Test: 18F-FGLN PET Imaging; Drug: (18F)FPGLU

INTERVENTIONS:
Diagnostic Test: 18F-FGLN PET Imaging — PET/CT Imaging: The study visit will take around 3-4 hours, the duration of PET will be around 90 minutes. Women should have negative pregnancy test prior to the study. An intravenous catheter will be placed in the subject's opposite arm, which will be used for radiotracer administration. A low-dose helical CT scan will be performed during a ~15 sec inspiratory breath hold and used for CT-based attenuation correction of PET emission data and as an anatomical reference for image analyses. Participants will be retained in the PET facility following the PET scan to promote urination to increase elimination of the radiotracer.
Drug: (18F)FPGLU — [F-18]FGln is a natural glutamine derivative was synthesized to explore its potential application of imaging glutamine uptake for cancer diagnosis. The proposed research study will provide preliminary evidence of the potential to utilize [F-18]FGln as a non-invasive imaging biomarker of glutamine flux and metabolism across a range of PAH subjects.

SUMMARY:
Pulmonary arterial hypertension (PAH) is mortal disease affecting the blood vessels of the lung. Despite its morbid prognosis, PAH is often misdiagnosed or ignored, with an average time of 44 months between onset of symptoms to diagnosis and substantial progression of disease severity. Therefore, a pressing need exists to develop non-invasive diagnostic imaging tools, particularly that can detect early disease stages.

Efforts have been made to develop such imaging capabilities through platform development of echocardiography, cardiac MRI, chest computed tomography (CT), and positron emission tomography (PET), among others. While some have demonstrated promise, few have shown a precise ability to offer disease quantifications of the diseased lung and vasculature itself, to detect early stages of disease, and to reflect alterations of the lung, vasculature, and right ventricle that reflect the molecular origins of this disease.

[F-18]FGln has been previously utilized in oncology studies as a non-invasive in vivo imaging biomarker of tumor glutamine flux and metabolism. Our preliminary in vivo pre-clinical rodent studies demonstrated that [F-18]FGln demonstrated increased uptake in diseased pulmonary vessels and the right ventricle in a rodent model of PAH. The proposed research study will provide preliminary evidence of the potential to utilize [F-18]FGln as a non-invasive imaging biomarker of glutamine flux and metabolism across a range of PAH subjects.

DETAILED DESCRIPTION:
Objective: Investigators will conduct in-human PET imaging of 18F-fluoroglutamine (18F-FGln) in patients with PAH to compare glutamine uptake to that of controls.

Specific Aim: Utilizing18F-FGln PET imaging to measure pathogenic glutamine uptake in patients with PAH or eiPAH and controls.

Significance: Investigator multi-disciplinary team, comprised of Drs. Chan, Tavakoli, and Mason are already actively collaborating together, and are uniquely positioned to image and quantify glutamine uptake in this special patient population. In doing so, investigators will determine the potential of this [F-18]FGln to serve as a non-invasive imaging biomarker of in vivo glutamine flux and metabolism associated with PAH Investigators are proposing a pilot experiment, Objective: Investigators will conduct in-human PET imaging of 18F-fluoroglutamine (18F-FGln) in patients with PAH to compare glutamine uptake to that of controls.

Specific Aim: Utilizing18F-FGln PET imaging to measure pathogenic glutamine uptake in patients with PAH or eiPAH and controls.

Significance: Investigator multi-disciplinary team, comprised of Drs. Chan, Tavakoli, and Mason are already actively collaborating together, and are uniquely positioned to image and quantify glutamine uptake in this special patient population. In doing so, investigators will determine the potential of this [F-18]FGln to serve as a non-invasive imaging biomarker of in vivo glutamine flux and metabolism associated with PAH

Investigators are proposing a pilot experiment, in which we will enroll the following subjects each group:

10 subjects with Idiopathic PAH (IPAH) 17 subjects with Scleroderma-PAH (SSc-PAH) 7 subjects with Scleroderma exercise induced PAH (SSc-eiPAH) 10 subjects with scleroderma but no PAH 27 healthy controls The cases will be matched for age/gender/race with 27 healthy controls for comparison.

If we had to recruit controls before cases, we will still be able to match cases and controls. We will initiate study visits with 1 or 2 controls, and matching 2 controls with 40 cases. 18F-FGN PET Imaging will be performed at The University of Pittsburgh's PET Research Facility.

Study visit: The study visit will take around 3-4 hours, the duration of PET scan will be around 90 minutes.

Upon subject arrival, CRC will do the following:

1. Review the medications the subject is currently on.
2. Take the subject vitals (Temperature/blood pressure/pulse).
3. Women of child-bearing potential (WCBP) will need to complete a urine pregnancy test on the day of the scan procedure, prior to any PET scan procedures. An intravenous catheter will be placed in the subject's arm, which will be used for radiotracer administration. All PET scans will be performed for a single bed position on a Siemens Biograph mCT Flow. Patients will be positioned in the scanner in a head-first supine orientation. A scout CT scan will be performed to fix the PET bed position such that the superior axial image planes are located approximately 1 cm above the lung apex, which will cover the axial extent of the heart and the majority of lung tissue. A low dose helical CT scan will be performed during a ~15 sec inspiratory breath hold and used for CT-based attenuation correction of PET emission data and as an anatomical reference for image analyses. Following the CT acquisition, approximately 10.0 mCi of 18F-FGln will be injected intravenously as a slow bolus (20 sec) and 90 minutes of PET emission data will be collected in list-mode. List-mode PET emission data will be binned into an ungated dynamic series of 28 frames for initial tracer kinetic analyses. Additional reconstructions will be performed with cardiac gating to isolate the end-diastole phase, respiratory gating to isolate the inspiratory respiratory phase, and dual gating (cardiac and respiratory gating) to achieve virtually motion-free PET images. These data will also be used to optimize reconstruction and gating parameters for future 18F-FGln studies.

If for reasons of participant discomfort or technical difficulty (problems with PET camera, cyclotron breakdown etc.), the full PET scanning procedure cannot be completed in 1 day we may be given the option to ask the participant to return within 30 days to complete the study. On this day, preparation will again consist of intravenous catheterization. The scanning protocol will be identical to that described above. Participant will not receive more than 2-3 CT scans and, no more than two [F-18] FGN PET scans with maximum effective dose exposure of 1.777 rads, as a result in participation in this research study. If participant had to be scheduled for a another day for this study, he/she will receive an additional IV line and will also have to undergo urine pregnancy testing (if applicable). Follow-up Procedures: A follow-up telephone call will be made to subjects by the research team approximately 1 to 7 days after the PET/CT scan to inquire about any adverse events the participant may have encountered related to the scans. Medical Record Information: We will request subjects' authorization to access medical record information from their past, current and future medical record information related to their health condition to be recorded into the Research study. This information will be collected from Heart and Vascular Institute (HVI) records, hospital records and, if applicable, private physician records. Since heart failure symptoms/progression may change over time, and these changes may be important to this study result, future medical records will be collected indefinitely. The medical record information contained within the study database will be used for research related purposes for an indefinite time. Subjects medical record information may be reviewed to see if they were eligible for any ongoing or future research studies; if they were eligible, then we may contact them

ELIGIBILITY:
Inclusion Criteria:

Cases:

1. Age between 18-75 years old
2. Confirmed diagnosis of SSc-PAH / SSc-eiPAH/IPAH/ by right heart catheterization. And Scleroderma with no PAH confirmand by echo.

Controls:

1. Age between 18-75 years old
2. Individuals who are at low risk for current or future cardiovascular or pulmonary symptoms or diseases

Exclusion Criteria:

Cases:

1. Smoking
2. Pregnant/ breast feeding women
3. Children under 18
4. Inability to read and understand the informed consent
5. History of CT contrast allergy
6. Inability to lie down for long period of time
7. Having claustrophobic
8. History of radiation exposure at workplace
9. Consuming more than 2-3 alcoholic drinks a week
10. Working previously in any of the following "cool miner, painter, iron miner, Mill worker, asbestos, insulation/heat resistance materials, sand"
11. Any medical conditions involving the heart or lungs that would make participation in the study unsafe in the opinion of the PI.

Controls:

1. Smoking
2. Pregnant/ breast feeding women
3. Children under 18
4. Inability to read and understand the informed consent
5. History of CT contrast allergy.
6. Inability to lie down for long period of time
7. Having claustrophobic
8. History of radiation exposure at workplace
9. Consuming more than 2-3 alcoholic drinks a week
10. Working previously in any of the following "coal miner, painter, iron miner, Mill worker, asbestos, insulation/heat resistance materials, sand"
11. Any medical conditions involving the heart or lungs or that would make participation in the study unsafe in the opinion of the PI.
12. Family history of Pulmonary Hypertension or Scleroderma

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Estimated)
Dates: Start 2022-07-11 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
SUV or image-based threshold of 18F-FGNnon-diseased controls | 90 minutes
  Regional [F-18] fluoroglutamine (18F-FGN) utilization will be measured as standardized uptake values (SUV) of 18F-FGN in right ventricle wall, left ventricle wall, and perivascular tissue within the lung parenchyma.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Chan, Principal Investigator — University of Pittsburgh
Locations (1):
- Montefiore Hospital Clinical and Translational Research Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data may be shared with other individuals for future research and if shared will be shared without identifiers.
  Participant's medical record information contained within the Research study may be provided to secondary research investigators (i.e., research investigators who are not affiliated with the Comprehensive Pulmonary Hypertension Program at University of Pittsburgh).The type of data shared would include demographic information, past medical history, medications, lab results, right heart Cath hemodynamics and cardiac imaging studies. However, prior to its provision to any secondary investigators, the information shall be de-identified. The Comprehensive Pulmonary Hypertension Program and Comprehensive lung center shall require secondary investigators to obtain regulatory approval prior its provision of de-identified information to the secondary investigators.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will available starting 6 months after publication
Access Criteria: The Comprehensive Pulmonary Hypertension Program and Comprehensive lung center shall require secondary investigators to obtain regulatory approval prior its provision of de-identified information to the secondary investigators